CLINICAL TRIAL: NCT01162070
Title: Uveitis: Medico-economical and Clinical Evaluation of a Standardized Strategy for an Etiological Diagnosis
Brief Title: Evaluation of a Standardized Strategy for Uveitis Etiological Diagnosis
Acronym: ULISSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009.566/19
Record Dates: First submitted 2010-07-12; First posted 2010-07-14 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Uveitis
Keywords: Uveitis; etiological diagnosis; standardized strategy
MeSH Terms: conditions — Uveitis | interventions — Bloodless Medical and Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Free strategy (Active Comparator): Free strategy followed in order to make the etiological diagnosis, which means, investigators are free to perform any examination they thought necessary.
  Interventions: Other: Free strategy
- Experimental strategy (Experimental): Etiological diagnosis made by following a standardized two-stage strategy: first-line assessment (listed examinations and then examinations directed by the clinical or para-clinical elements of orientation) and second or third-line assessment (examinations directed by the anatomo-clinical type of uveitis).
  Interventions: Other: Standardized strategy

INTERVENTIONS:
Other: Free strategy — Free strategy followed in order to make the etiological diagnosis, which means, investigators are free to perform any examination they thought necessary.
  Other Names: Procedure or strategy leading to the etiological diagnosis of the uveitis.
  Arms: Free strategy
Other: Standardized strategy — Etiological diagnosis made by following a standardized two-stage strategy: first-line assessment (listed examinations and then examinations directed by the clinical or para-clinical elements of orientation) and second or third-line assessment (examinations directed by the anatomo-clinical type of uveitis).
  Arms: Experimental strategy

SUMMARY:
The Uveitis, the inflammation of the uvea, is a rare disease with an incidence of 52/100,000 inhabitants per year and a prevalence of 115 / 100,000 inhabitants per year.

The causes of uveitis are numerous and include infectious diseases, systemic and neurological diseases, ophthalmic entities, neoplasia, and drug-related reactions. The etiological diagnosis is important both for prognosis and therapeutics.

However, clinical evaluations to establish etiological diagnosis are not standardized. Some authors suggest a minimalist examination, common to all kinds of uveitis. On the other hand, others propose an evaluation guided by the anatomo-clinical type of uveitis.

We conducted a retrospective study to assess the contribution of complementary examinations to etiological determination. In this study, we found that most patients benefited from a wide paraclinical evaluation compared to what is usually described in the literature. Complementary examinations were mostly systematic, without any clinical or ophthalmological elements of orientation. This study highlighted the lack of contribution of some examinations.

Using these results, and the literature analysis, we designed a diagnostic algorithm adapted to the anatomo-clinical type of uveitis.

Moreover, we found that the average cost per patient was estimated at €290.51 with the algorithm compared to €560.83 without it.

We would like to carry out a new study to estimate the efficiency as well as the medico-economic impact of the use of a standardized strategy for the etiological diagnosis of uveitis, compared with a free strategy.

Hypothesis:

* The standardized strategy for the diagnostic of uveitis is at least as efficient as the free one, and costs half as much.
* The examinations prescribed, except for those from the standardized strategy, do not contribute to etiological determination.

ELIGIBILITY:
Inclusion Criteria:

* Uveitis
* Patient consulting one of the study's sites
* Age > 18 years old
* Affiliation to the French national health insurance program
* Patient agreeing to participate in the study

Exclusion Criteria:

* Positive HIV serology
* Postsurgical or posttraumatic uveitis or endophthalmitis
* Toxoplasmic uveitis
* Pathology likely to be the cause of the known uveitis
* Ophthalmic entities only diagnosed by the ophthalmic examination
* Age < 18 years old
* Patient under law protection or guardianship
* Pregnant women or those planning to be pregnant during the study
* Severe uveitis (VA < 20/200) with retinal vascularitis requiring an emergency treatment and assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 905 (Actual)
Dates: Start 2010-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the percentage of patients having an etiological diagnosis 6 months after the beginning of the study for both strategies. | 6 months
  Note: Only diagnoses made at the end of the standardized strategy will be numbered in this arm of the study; all diagnoses made after by the free authorized examinations in this same arm will lead to standardized strategy failure.

SECONDARY OUTCOMES:
Clinical criteria concerning the standardized strategy | 6 months
  * Percentage of patients having an established etiological diagnosis at the end of the first diagnostic stage and at the end of the second diagnostic stage. (Second or third-line assessment).
  * Ratio of the standardized strategy's first stage examinations having contributed to the etiological diagnosis.
  * Ratio of the standardized strategy's second stage examinations, directed by the anatomo-clinical type of the uveitis (Second or third-line assessment) having contributed to an etiological diagnosis.
  * Ratio of free complementary examinations having contributed to an etiological diagnosis.
Clinical criteria concerning the free strategy | 6 months
  * Description and ratio of the examinations that have not allowed the doctor to make an etiological diagnosis.
  * Description and ratio of the complementary examinations not included in the standardized strategy.
The average cost of economic criteria for each strategy. | 12 months
  * For each patient: The standardized strategy's average cost of diagnosis distinguishing between first diagnostic stage costs and second diagnostic stage costs (made up of the second or third-line assessment directed by the anotomo-clinical type of the uveitis).
  * Average cost of the complementary examinations not included in the standardized strategy but allowed at the end of it (subsequent free assessment).
  * Average cost for each patient of the whole free strategy.
Quality of life criteria | : 6 months
  - Quality of life, estimated with the standard quality of life questionnaire (SF-36) and the one specific to ophthalmology (NEI VFQ-25), will be compared between these groups:
  1. Uveitis diagnosis versus no diagnosis
  2. Free strategy versus standardized strategy.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Médecine Interne, Hospices Civils de Lyon (HCL)-Hôpital de la Croix Rousse, Lyon, France

REFERENCES:
- [Background] de Parisot A, Kodjikian L, Errera MH, Sedira N, Heron E, Perard L, Cornut PL, Schneider C, Riviere S, Olle P, Pugnet G, Cathebras P, Manoli P, Bodaghi B, Saadoun D, Baillif S, Tieulie N, Andre M, Chiambaretta F, Bonin N, Bielefeld P, Bron A, Mouriaux F, Bienvenu B, Vicente S, Bin S, Broussolle C, Decullier E, Seve P; ULISSE group. Randomized Controlled Trial Evaluating a Standardized Strategy for Uveitis Etiologic Diagnosis (ULISSE). Am J Ophthalmol. 2017 Jun;178:176-185. doi: 10.1016/j.ajo.2017.03.029. Epub 2017 Mar 31. PMID 28366648